CLINICAL TRIAL: NCT05409053
Title: Open Reduction and Kirschner Wires Fixation Versus Cannulated Screws Internal Fixation for Displaced Lateral Condyle Humeral Fracture in Children. Randomized Controlled Trial.
Brief Title: Kirschner Wires Fixation Versus Cannulated Screws Internal Fixation for Displaced Lateral Condyle Humeral Fracture in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Bassam Abdelrahim Abdelbasset, resident doctor at orthopaedic department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: soh-Med-22-03-08
Record Dates: First submitted 2022-03-16; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Lateral Condyle Humerus Fracture in Children
MeSH Terms: interventions — Open Fracture Reduction; Closed Fracture Reduction; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- screw fixation (Active Comparator): lateral condyle humerus fracture open reduction and internal fixation by canullated screws
  Interventions: Procedure: open reduction
- k wire fixation (Active Comparator): lateral condyle humerus fracture open reduction and internal fixation by K wire
  Interventions: Procedure: open reduction
- Conservative management (Other): Undisplaced fractured treated conservatively by above elbow slab
  Interventions: Other: Conservative management
- Closed reduction and percutaneous pinning (Other): Undisplaced fractured treated closed reduction and percutaneous pinning
  Interventions: Procedure: Closed reduction

INTERVENTIONS:
Procedure: open reduction — the displaced fractures will be treated with open reduction so as to achieve the near anatomical alignment
  Arms: k wire fixation; screw fixation
Procedure: Closed reduction — the non displaced fractures will be treated with closed reduction and percutaneous pinning
  Arms: Closed reduction and percutaneous pinning
Other: Conservative management — the non displaced fractures will be treated with closed reduction and castor slab
  Arms: Conservative management

SUMMARY:
Lateral condyle fracture of the distal humerus is the second most common injury around the elbow and accounts for 20% of all the elbow fractures in children.The average age for the fracture involving the lateral condyle is around six years.

There are different treatment options of the lateral condyle fractures include

* non-operative management with plaster cast immobilization for undisplaced or minimally displaced fractures.
* Whereas the fractures displaced >2 mm need operative management. The objective of treatment in the displaced fracture is to obtain and maintain the articular congruity.

In the operative management, the reduction technique includes open or closed methods.

ELIGIBILITY:
Inclusion Criteria:

* Children up to 14 years.
* closed lateral condylar fracture.
* displacement more than 2mm .
* fracture Less than two weeks of injury.

Exclusion Criteria:

* Patients with open fractures.
* otherassociated injury in the same elbow .
* elbow with preexisting anatomical deformity .

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Time of union | 6 Months
  Follow up radiographs will be requested at immediate postoperative 2, 4, 6, 12 and 24 weeks postoperative to assess healing

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Franks D, Shatrov J, Symes M, Little DG, Cheng TL. Cannulated screw versus Kirschner-wire fixation for Milch II lateral condyle fractures in a paediatric sawbone model: a biomechanical comparison. J Child Orthop. 2018 Feb 1;12(1):29-35. doi: 10.1302/1863-2548.12.170090. PMID 29456751
- [Background] Justus C, Haruno LS, Riordan MK, Wilsford L, Smith T, Antekeier S, McKay SD. Closed and Open Reduction of Displaced Pediatric Lateral Condyle Humeral Fractures, a Study of Short-Term Complications and Postoperative Protocols. Iowa Orthop J. 2017;37:163-169. PMID 28852352
- [Background] Cardona JI, Riddle E, Kumar SJ. Displaced fractures of the lateral humeral condyle: criteria for implant removal. J Pediatr Orthop. 2002 Mar-Apr;22(2):194-7. PMID 11856929
- [Background] Baharuddin M, Sharaf I. Screw osteosynthesis in the treatment of fracture lateral humeral condyle in children. Med J Malaysia. 2001 Dec;56 Suppl D:45-7. PMID 14569766